CLINICAL TRIAL: NCT04389086
Title: Multicentre, Open-label, Randomised, Controlled, Parallel Arms Clinical Trial of Induction Chemotherapy Followed by Chemoradiotherapy Versus Chemoradiotherapy Alone as Neoadjuvant Treatment for Locally Recurrent Rectal Cancer - PelvEx II
Brief Title: Induction Chemotherapy for Locally Recurrent Rectal Cancer
Acronym: PelvEx II
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Principal Investigator, J. W. A. Burger, MD, PhD, Catharina Ziekenhuis Eindhoven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL73593
Record Dates: First submitted 2020-05-07; First posted 2020-05-15 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-09

CONDITIONS: Recurrent Rectal Cancer
Keywords: Locally recurrent rectal cancer; Neoadjuvant therapy; Induction chemotherapy; Resection margin
MeSH Terms: conditions — Rectal Neoplasms; Margins of Excision | interventions — Drug Combinations; Folfox protocol; IFL protocol; Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Induction chemotherapy + chemoradiotherapy + surgery (Experimental): Induction chemotherapy followed by neoadjuvant chemoradiotherapy and surgery
  Interventions: Drug: Combination drug; Radiation: Chemoradiotherapy; Procedure: Surgery locally recurrent rectal cancer
- Neoadjuvant chemotherapy + surgery (Active Comparator): Neoadjuvant chemoradiotherapy followed by surgery
  Interventions: Radiation: Chemoradiotherapy; Procedure: Surgery locally recurrent rectal cancer

INTERVENTIONS:
Drug: Combination drug — Induction chemotherapy consists of either three three-weekly cycles of CAPOX (oxaliplatin 130 mg/m2 BSA IV + capecitabine 1000 mg/m2 BSA, orally, twice daily) or four two-weekly cycles of FOLFOX (85 mg/m2 BSA of oxaliplatin IV + 400 mg/m2 BSA of leucovorin IV + 400 mg/m2 BSA of bolus 5-fluorouracil IV followed by 2400 mg/m2 BSA of continuous 5-fluorouracil IV). It is left to the discretion of the treating medical oncologist which of the two will be administered. In case of (previous) unacceptable toxicity (physician's discretion) to oxaliplatin, FOLFIRI may be prescribed. FOLFIRI (180 mg/m2 BSA of irinotecan IV + 400 mg/m2 BSA of leucovorin IV + 400 mg/m2 BSA of bolus 5-fluorouracil IV followed by 2400 mg/m2 BSA of continuous 5-fluorouracil IV) consists of four two-weekly cycles.
  If a patient has stable or responsive disease, induction chemotherapy will be continued with either one three-weekly cycle of CAPOX or two two-weekly cycles of FOLFOX/FOLFIRI.
  Other Names: CAPOX; FOLFOX; FOLFIRI
  Arms: Induction chemotherapy + chemoradiotherapy + surgery
Radiation: Chemoradiotherapy — Concomitant chemotherapy agent: capecitabine
  Radiotherapy dose: full course radiotherapy consists of 25x2.0 or 28x1.8 Gy. In case of previous radiotherapy, the radiotherapy dose will consist of 15x2.0 Gy.
Procedure: Surgery locally recurrent rectal cancer — Type of surgery depends on the location of the recurrence and involvement of adjacent structures and is left to the discretion of the operating surgeon.
  Intraoperative radiotherapy is optional.

SUMMARY:
This is a multicentre, open-label, parallel arms, phase IIII study that randomises patients with locally recurrent rectal cancer in a 1:1 ratio to receive either induction chemotherapy followed by neoadjuvant chemoradiotherapy and surgery (experimental arm) or neoadjuvant chemoradiotherapy and surgery alone (control arm)

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Confirmed locally recurrent rectal cancer after total or partial mesorectal resection for rectal or distal sigmoidal cancer either by histopathology ór clinically proven (evidence on imaging in combination with clinical findings, with consensus in MDT)
* Resectable disease determined by magnetic resonance imaging (MRI) or deemed resectable after neoadjuvant treatment with chemoradiotherapy.
* WHO performance score 0-1
* Written informed consent

Exclusion Criteria:

* Radiological evidence of metastatic disease (e.g. liver, lung) at time of randomisation or in the six months prior to randomisation.
* Known homozygous DPD deficiency
* Any chemotherapy in the past 6 months.
* Any contraindication for the planned chemotherapy, as determined by the medical oncologist.
* Radiotherapy in the past 6 months for primary rectal cancer.
* Any contraindication for the planned chemoradiotherapy, as determined by the medical oncologist and/or radiation oncologist.
* Any contraindication for surgery, as determined by the surgeon and/or anaesthesiologist.
* Concurrent malignancies that interfere with the planned study treatment or the prognosis of resected LRRC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 364 (Estimated)
Dates: Start 2020-11-13 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2030-03-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with a clear resection margin | Scored within 1 one month of surgery
  A resection margin is considered clear (R0), if there are no tumour cells in any of the resection surfaces as determined by microscopy (resection margin > 0mm)

SECONDARY OUTCOMES:
Local recurrence free survival | Assessed up to 5 years
Progression free survival | Assessed up to 5 years
Metastasis free survival | Assessed up to 5 years
Disease free survival | Assessed up to 5 years
Overall survival | Assessed up to 5 years
Pathologic response | Scored within 1 month of surgery
  Scored according to Mandard
Toxicity induction chemotherapy | Scored until one month after the last administration of the chemotherapy
  Adverse events grade 3 or higher according to the NCI-CTCAE v5.0
Compliance induction chemotherapy | Scored within 1 month after start chemoradiotherapy
Toxicity chemoradiotherapy | Scored until 3 months after the last administration of the radiotherapy
  Adverse events grade 3 or higher according to the NCI-CTCAE v5.0
Compliance chemoradiotherapy | Evaluation at time of surgery
Number of patients undergoing surgery | Surgery is scheduled 10-14 weeks after finishing chemoradiotherapy
Surgical characteristics | Evaluation directly postoperative
  including data on intra-operative radiotherapy
Major surgical morbidity | 30 and 90-days postoperative
  Clavien-Dindo grade 3 or higher
Radiological response | Restaging is performed after 3 cycles of CAPOX (1 cycle is 3 weeks) or 4 cycles of CAPOX/FOLFOX (1 cycle is 2 weeks). Second restaging is performed 4-6 weeks after finishing chemoradiotherapy
  mrTRG
Cancer specific quality of life | at baseline, 3 months and 12 months postoperative
  QLQ-C30
Cost-effectiveness | at baseline, 3 months and 12 months postoperative
  EQ-5D-5L
Colorectal cancer specific quality of life | at baseline, 3 months and 12 months postoperative
  QLQ-CR29

CONTACTS AND LOCATIONS:
Overall Officials: Pim Burger, MD, Principal Investigator — Catharina Ziekenhuis Eindhoven
Locations (14):
- UZ Gent, Ghent, Belgium
- Netherlands (8):
  - Amsterdam UMC, Amsterdam
  - Antoni van Leeuwenhoek, Amsterdam
  - Catharina Hospital, Eindhoven
  - University Medical Centre Groningen, Groningen
  - Leids University Medical Centre, Leiden
  - Haaglanden Medical Centre, Leidschendam
  - Maastricht University Medical Centre, Maastricht
  - Erasmus Medical Centre, Rotterdam
- Oslo Universitetssykehus, Oslo, Norway
- Instituto Portugues de Oncologia de Lisboa Francisco Gentil, E.P.E., Lisbon, Portugal
- Sweden (3):
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Skåne Universitetssjukhuset, Malmo
  - Karolinska Universitetssjukhuset, Stockholm

IPD SHARING:
Plan to Share IPD: Yes
Participant-level datasets and statistical codes will become available upon reasonable request after the results of the study have been published.
Supporting Information: Study Protocol, ICF
Time Frame: The full protocol and Dutch informed consent forms are publicly accessible after approval of the medical ethics committee.